CLINICAL TRIAL: NCT02037594
Title: Intervention to Enhance PrEP Uptake and Adherence in a Community-Based Setting
Acronym: SPARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Sarit Golub, Associate Professor, Hunter College of City University of New York
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 349555-6; R01AA022067 (NIH)
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Human Immunodeficiency Virus (HIV)
Keywords: HIV; Pre-exposure prophylaxis; PrEP; MSM; Demonstration Project
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Counseling + SOC Adherence (Experimental): Sexual Health Counseling followed by Standard of Care Adherence Support
  Interventions: Behavioral: Sexual Health Counseling; Behavioral: Standard of Care Adherence Support (Active Control)
- Counseling + Enhanced Adherence (Experimental): Sexual Health Counseling followed by Enhanced Adherence Intervention
  Interventions: Behavioral: Sexual Health Counseling; Behavioral: Enhanced Adherence Intervention
- Information + SOC Adherence (Experimental): PrEP Information followed by Standard of Care Adherence Support
  Interventions: Behavioral: PrEP Information (Active Control); Behavioral: Standard of Care Adherence Support (Active Control)
- Information + Enhanced Adherence (Experimental): PrEP Information followed by Enhanced Adherence Intervention
  Interventions: Behavioral: Enhanced Adherence Intervention; Behavioral: PrEP Information (Active Control)

INTERVENTIONS:
Behavioral: Sexual Health Counseling — This brief intervention presents PrEP within the context of a patient's comprehensive sexual health plan and is designed to enhance decision-making around PrEP use and decrease sexual risk taking.
  Arms: Counseling + Enhanced Adherence; Counseling + SOC Adherence
Behavioral: Enhanced Adherence Intervention — This brief intervention is provides standard of care PrEP adherence information plus specific counseling, troubleshooting, and support.
  Arms: Counseling + Enhanced Adherence; Information + Enhanced Adherence
Behavioral: PrEP Information (Active Control) — Standard of Care Information about PrEP
  Arms: Information + Enhanced Adherence; Information + SOC Adherence
Behavioral: Standard of Care Adherence Support (Active Control) — Standard of care information and instruction about PrEP adherence.
  Arms: Counseling + SOC Adherence; Information + SOC Adherence

SUMMARY:
This study identifies social and behavioral factors likely to influence PrEP acceptability and adherence among men who have sex with men (MSM), and collaborates with a community health center to evaluate a two-stage intervention to improve PrEP decision-making, as well as persistence and adherence for those who chose to take PrEP.

DETAILED DESCRIPTION:
Pre-exposure prophylaxis (PrEP) refers to daily or intermittent oral administration of antiretroviral drugs designed to protect high-risk HIV-negative individuals from infection. In order for PrEP to become an effective prevention tool, three critical factors must be addressed: a) acceptability, i.e., individuals who would benefit from PrEP must know about it and be willing to take it; b) adherence, i.e., individuals who choose to PrEP as a prevention strategy must take the pills as prescribed; and c) implementation, i.e., processes and protocols must be developed to allow for the integration of PrEP delivery and programs into real world settings in a way that is feasible, scalable, and realistic. This project has three specific aims: 1) Identifying social and behavioral factors that are likely to influence PrEP implementation, acceptance, and use/adherence by men who have sex with men (MSM) in NYC, including factors at individual-, community-, and organizational-levels; 2) Examining social and behavioral factors associated with disparities in access to prevention and care services among MSM in NYC that might directly impact PrEP implementation programs and policies; and 3) Evaluating an intervention in which PrEP is introduced, provided, and supported as part of a prevention package delivered in an community health center. The project has the potential to exert a sustained and powerful influence not only on the effectiveness of PrEP interventions for MSM, but also on dissemination and scalability of a targeted intervention within community-based settings and in a manner that reduces disparities in access and maximizes cultural competence and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Registered patient receiving medical or health services at Callen-Lorde Community Health Center
* Male sex (at birth) and reported sex with men or transwomen
* At least 18 years of age
* HIV-negative
* At risk for HIV acquisition

Exclusion Criteria:

* Past history of PrEP use or currently taking PrEP

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2014-01-30 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
PrEP Uptake | BL through 3-months
  Whether or not the patient decides to take PrEP
PrEP Persistence | BL through 12-months
  Whether or not patients who decide to take PrEP persist with the medication for the duration of the study.
PrEP Adherence | BL through 12 months
  Biological measure of medication adherence using dried blood spots, and self-report measure of adherence using VAS.
Sexual Risk Behavior | BL through 12-months
  Measured through STI testing and self-report.

CONTACTS AND LOCATIONS:
Overall Officials: Sarit A Golub, PhD, MPH, Principal Investigator — Hunter College, CUNY
Locations (1):
- Callen-Lorde Community Health Center, New York, New York, United States

REFERENCES:
- See also: Study Website — http://www.cunyhart.org/spark